CLINICAL TRIAL: NCT01912313
Title: Measuring Nerve Activity in Small Human Intestinal Biopsies in IBS (Irritable Bowel Syndrome)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Guy Boeckxstaens, Prof. Dr., KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: S55484
Record Dates: First submitted 2013-07-29; First posted 2013-07-31 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: IBS; Healthy
Keywords: IBS patients; healthy subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rectal biopsy (Experimental)
  Interventions: Procedure: Rectal biopsies from IBS patients or healthy subjects will be taken during proctoscopy

INTERVENTIONS:
Procedure: Rectal biopsies from IBS patients or healthy subjects will be taken during proctoscopy

SUMMARY:
Rectal biopsies from IBS patients or healthy subjects will be taken.

Biopsies will be used for:

1. the isolation of submucosal plexus to perform: 1.1 live nerve recordings and Calcium imaging; 1.2 immunohistochemistry; 1.3 mRNA (Messenger ribonucleic acids) isolation and real time PCR (Polymerase chain reaction);
2. culturing biopsies

On the basis of these observations, the general aim of the study is to move a significant step forward in the current knowledge on human ENS (enteric nervous system) in IBS by establishing a live imaging method to record enteric nerves activity in small intestinal biopsies from humans. This development is unique in its kind as not other research groups have reported successful live recordings with calcium imaging in this preparation.

In particular, the investigators aim:

1. to develop and validate the technique to measure activity in human enteric nerves in the submucous plexus isolated from rectal biopsies from healthy subjects and IBS patients;
2. to characterize this nerve activity in healthy subjects and IBS patients using both calcium imaging to evaluate the effect of different neuromodulators, immunohistochemistry and rtPCR to determine receptor expression levels and identify neurons and glial cells in the submucous ganglia;
3. to investigate whether the biopsies of IBS patients secrete more modulators/cytokines compared to healthy subjects and their potential to activate neurons.
4. to evaluate the influence of different food constituents (cow"s milk, wheat, yeast, gluten and soy) on the local reaction of the rectal mucosa and evaluate mast cell activation/degranulation in biopsies of IBS patients compared to healthy subjects.
5. To evaluate the amount of inflammatory mediators/metabolites in urine samples of IBS patients and healthy volunteers by the use of metabolic profiling

ELIGIBILITY:
Inclusion Criteria:

* IBS patients (based on ROME III Criteria)
* Healthy subjects

Exclusion Criteria:

- All subjects with not IBS related complaints

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99999999 (Estimated)
Dates: Start 2013-08; Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
nerve activity in healthy subjects and IBS patients | Starting from the moment biopsies are collected untill nerve activity in samples is lost (approximately 5 hours)
  Measuring nerve activity in healthy subjects and IBS patients using both calcium imaging to evaluate the effect of different neuromodulators, immunohistochemistry and rtPCR to determine receptor expression levels and identify neurons and glial cells in the submucous ganglia.

CONTACTS AND LOCATIONS:
Overall Officials: Guy Boeckxstaens, MD, Principal Investigator — Catholic University Leuven and Universitary Hospitals Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Vlaams-Brabant, Belgium